CLINICAL TRIAL: NCT02990949
Title: The Impact of the Timing of Trigger on IVF Success: Randomized Control Trial
Brief Title: The Impact of the Timing of Trigger on IVF Success
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to lack of enrollement
Sponsor: Colorado Center for Reproductive Medicine (Other)
Collaborators: Fertility Laboratories Of Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160397
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Fertilization in Vitro; Infertility; Embryonic Development
MeSH Terms: conditions — Infertility

ARMS (2):
- Testing group (Experimental): Timing of trigger at end of ovarian stimulation in an IVF cycle: trigger when 2 follicles reach 18mm, OR 1 follicle reaches 18mm AND 1 follicle is between 16-18mm.
  Interventions: Other: Timing of trigger
- Control group (No Intervention)

INTERVENTIONS:
Other: Timing of trigger
  Arms: Testing group

SUMMARY:
The aim of this study is to examine the length of ovarian stimulation with the timing of trigger in an IVF cycle and its potential to impact patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Planning to move forward with an IVF cycle
* Have met the requirements of being a patient at CCRM Colorado
* AMA: 39-44 years old And/or
* DOR: AMH < 1 & FSH >10 (age independent)

Exclusion Criteria:

* Contraindication for pregnancy
* Have not fulfilled requirements for IVF cycle
* Single gene couple or chromosomal rearrangement
* Severe male factor or testicular surgical sperm removal (need sufficient sperm for ICSI)
* One ovary
* Uterine anomalies
* Stage III or IV endometriosis
* Explained recurrent miscarriage
* PCO or PCOS
* Using donor oocyte or gestational carrier

Ages: 26 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Euploid Embryos: the percentage of euploid embryos produced as analyzed by comprehensive chromosomal screening, of total embryos tested | 4 weeks after egg retrieval

SECONDARY OUTCOMES:
Egg maturation: the proportion of mature eggs of total number of eggs retrieved | 1 week after egg retrieval
Live birth outcomes: the incidence of pregnancy resulting in live birth following embryo transfer of embryos produced by this IVF cycle | 9 months after frozen embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Katz-Jaffe, PhD, Study Director — CCRM, FLC
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States